CLINICAL TRIAL: NCT01836432
Title: A Phase III Study of Chemotherapy With or Without Algenpantucel-L (HyperAcute®-Pancreas) Immunotherapy in Subjects With Borderline Resectable or Locally Advanced Unresectable Pancreatic Cancer
Brief Title: Immunotherapy Study in Borderline Resectable or Locally Advanced Unresectable Pancreatic Cancer
Acronym: PILLAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG0505; 1210-1195 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer; Pancreatic Carcinoma Non-resectable; Locally Advanced Malignant Neoplasm
Keywords: Pancreatic Cancer; Immunotherapy; Vaccine Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Gemcitabine; Capecitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FOLFIRINOX + Algenpantucel-L (HAPa) Immunotherapy (Experimental): Arm 1A: SOC FOLFIRINOX + Algenpantucel-L (HAPa) Immunotherapy
  Day 71-80 Disease evaluated: New distant disease = salvage regimen Gem/Nab-Paclitaxel (6 cycles) + HAPa given days 8 and 22 for up to 18 doses total.
  Day 71-80 Disease evaluated: No distant disease = 5-FU or capecitabine plus Radiation+ HAPa on days 1 and 15 of Chemoradiotherapy.
  Post-Chemoradiation Disease evaluation: surgically resectable = surgery + adjuvant SOC Gemcitabine + HAPa given 1 and 15 for up to 18 doses total.
  Post-Chemoradiation Disease evaluation: not eligible for surgical resection (Stable) = continue FOLFIRINOX bi-weekly + HAPa bi-weekly 7 days offset from FOLFIRINOX up to18 doses of algenpantucel-L Immunotherapy.
  Post-Chemoradiation Disease evaluation: non-eligible for surgical resection (Progression) = salvage Gem/Nab-Paclitaxel (6 cycles) + HAPa given days 8 and 22 for up to 18 doses total.
  Interventions: Drug: FOLFIRINOX; Biological: Algenpantucel-L Immunotherapy; Radiation: 5-FU Chemoradiation; Drug: Gemcitabine; Drug: Capecitabine; Drug: Nab-Paclitaxel
- FOLFIRINOX (SOC) ALONE (Active Comparator): Arm 2A: FOLFIRINOX (Oxaliplatin 85 mg/m^2 IV over 2 hours; Irinotecan 180 mg/m^2 IV over 90 minutes; Leucovorin 400 mg/m^2 IV over 2 hours; Fluorouracil 2.4 g/m^2 IV over 46 hours) given days 1, 15, 29, 43 & 57
  Day 71-80 Disease eval: New disease = salvage Gem/Nab-Paclitaxel: nab-paclitaxel 125mg/m^2 IV over 30-40 minutes followed by gemcitabine 1000 mg/m^2 IV over 30-60 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest
  Day 71-80 Disease eval: No disease = 5-FU or capecitabine plus Radiation (5-FU continuous IV infusion of 200-250 mg/m^2/day given 5-7 days each week over 5.5 weeks or Capecitabine 825 mg/m^2 PO BID M-F) concurrently with external beam radiation given at 1.8 Gy per fraction for 28 fractions total dose of 50.4 Gy
  Post-XRT Disease eval: surgically resectable = surgery + adjuvant SOC Gemcitabine
  Ineligible for surgical resection & stable disease = continue FOLFIRINOX
  Ineligible for surgical resection & progressive disease = salvage Gem/Nab-Paclitaxel
  Interventions: Drug: FOLFIRINOX; Radiation: 5-FU Chemoradiation; Drug: Gemcitabine; Drug: Capecitabine; Drug: Nab-Paclitaxel
- Gemcitabine/Nab-Paclitaxel+Algenpantucel-L HAPa Immunotherapy (Experimental): Arm 1B: Gemcitabine/Nab-Paclitaxel + Algenpantucel-L (HAPa) Immunotherapy
  Day 71-80 Disease evaluated: New distant disease = salvage regimen FOLFIRINOX + HAPa given every 14 days (alternate weeks of FOLFIRINOX) for up to 18 doses total.
  Day 71-80 Disease evaluated: No distant disease = 5-FU or capecitabine plus Radiation + HAPa on days 1 and 15 of Chemoradiotherapy.
  Post-Chemoradiation Disease evaluation: surgically resectable = surgery + adjuvant SOC Gemcitabine + HAPa given days 1 and 15 for up to 18 doses total.
  Post-Chemoradiation Disease evaluation: not eligible for surgical resection (Stable) = continue Gem/Nab-Paclitaxel + HAPa given on days 8 and 22 for up to18 doses of algenpantucel-L Immunotherapy.
  Post-Chemoradiation Disease evaluation: non-eligible for surgical resection (Progression) = salvage FOLFIRINOX + HAPa given every 14 days (alternate weeks of FOLFIRINOX) for up to 18 doses total.
  Interventions: Drug: FOLFIRINOX; Biological: Algenpantucel-L Immunotherapy; Radiation: 5-FU Chemoradiation; Drug: Gemcitabine; Drug: Capecitabine; Drug: Nab-Paclitaxel
- Gemcitabine/Nab-Paclitaxel (SOC) Alone (Active Comparator): Arm 2B: Gemcitabine/Nab-Paclitaxel (SOC) Alone
  SOC Gem/Nab-Paclitaxel: nab-paclitaxel 125mg/m^2 IV over 30-40 minutes followed by gemcitabine 1000 mg/m^2 IV over 30-60 minutes for 3 weeks with 1 week rest. Given on days 1, 8, 15, 29, 36, 43, 57, 64 and 71
  Day 71-80 Disease evaluated: New distant disease = salvage FOLFIRINOX given every 14 days
  Day 71-80 Disease evaluation: No disease = 5-FU or capecitabine plus Radiation (5-FU continuous IV infusion of 200-250 mg/m^2/day given 5-7 days each week over 5.5 weeks or Capecitabine 825 mg/m^2 PO BID M-F) concurrently with external beam radiation given at 1.8 Gy per fraction for 28 fractions total dose of 50.4 Gy
  Post-XRT Disease eval: surgically resectable = surgery + adjuvant SOC Gemcitabine
  Ineligible for surgical resection & stable disease = continue gem/nab-paclitaxel given for 3 weeks (days 1, 8 and 15) with 1 week rest
  Ineligible for surgical resection & progressive disease = salvage FOLFIRINOX given every 14 days
  Interventions: Drug: FOLFIRINOX; Radiation: 5-FU Chemoradiation; Drug: Gemcitabine; Drug: Capecitabine; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: FOLFIRINOX — FOLFIRINOX consisting of Oxaliplatin 85 mg/m^2 IV over 2 hours; Irinotecan 180 mg/m^2 IV over 90 minutes; Leucovorin 400 mg/m^2 IV over 2 hours; Fluorouracil 2.4 g/m^2 IV over 46 hours
  Other Names: Oxaliplatin; Eloxatin®; Irinotecan; Camptosar®; Leucovorin; Citrovorum factor; folinic acid; Fluorouracil; 5-Fluorouracil; 5-FU
Biological: Algenpantucel-L Immunotherapy — Algenpantucel-L Immunotherapy (HAPa) consisting of 300 Million HAPa cells given by intradermal injection
  Other Names: HyperAcute®-Pancreas; HAPa
  Arms: FOLFIRINOX + Algenpantucel-L (HAPa) Immunotherapy; Gemcitabine/Nab-Paclitaxel+Algenpantucel-L HAPa Immunotherapy
Radiation: 5-FU Chemoradiation — 5-FU Chemoradiation consisting of 5-FU continuous IV infusion of 200-250 mg/m^2/day given 5-7 days each week over 5.5 weeks concurrently with external beam radiation
  Other Names: Fluorouracil; 5-Fluorouracil; 5-FU
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 given intravenously over 30 minutes for 3 weeks (days 1, 8 and 15) with 1 week rest.
  Other Names: Gemzar
Drug: Capecitabine — Capecitabine consisting of 825 mg/m^2 PO BID M-F concurrently with external beam radiation
  Other Names: Xeloda
Drug: Nab-Paclitaxel — Nab-Paclitaxel 125 mg/m^2 given intravenously over 30-40 minutes
  Other Names: Abraxane; Paclitaxel

SUMMARY:
Unfortunately, despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with pancreatic cancer continue to die from the rapid progression of their disease. One primary reason for this is that the disease is typically without symptoms until significant local and/or distant spread has occurred and is often beyond the chance for cure at the time of the diagnosis. The lack of any treatment to substantially increase long term survival rates is reflected by the poor outcomes associated with this disease, specifically time to disease progression and overall survival.

However, another important part of the body is now being looked at as a target for therapy against this disease - the immune system. Scientists have clearly shown that pancreatic tumor cells produce a number of defective proteins, or express normal proteins in highly uncharacteristic ways, as part of this cancer. In some cancers, these abnormalities can cause an immune response to the cancer cells much in the way one responds to infected tissue. In progressive cancers however, the immune system fails to effectively identify or respond to these abnormalities and the cancer cells are not attacked or destroyed for reasons not yet fully understood. This clinical trial proposes a new way to stimulate the immune system to recognize pancreatic cancer cells and to stimulate an immune response that destroys or blocks the growth of the cancer.

This new method of treatment helps the immune system of pancreatic cancer patients to "identify" the cancerous tissue so that it can be eliminated from the body. As an example, most people are aware that patients with certain diseases may require an organ transplant to replace a damaged kidney or heart. After receiving their transplant, these patients receive special drugs because they are at great danger of having an immune response that destroys or "rejects" the transplanted organ. This "rejection" occurs when their immune system responds to differences between the cells of the transplanted organ and their own immune system by attacking the foreign tissue in the same way as it would attack infected tissue. When the differences between foreign tissues and the patient's body are even larger, as with the differences between organs from different species, the rejection is very rapid, highly destructive, and the immunity it generates is longlasting. This is called hyperacute rejection and the medicine used to immunize patients in this protocol tries to harness this response to teach a patient's immune system to fight their pancreatic cancer just as the body would learn to reject a transplanted organ from an animal.

To do this, Algenpantucel-L immunotherapy contains human pancreatic cancer cells that contain a mouse gene that marks the cancer cells as foreign to patient's immune systems. The immune system therefore attacks these cancer cells just as they would attack any truly foreign tissue, destroying as much as it can. Additionally, the immune system is stimulated to identify differences (aside from the mouse gene) between these cancer cells and normal human tissue as foreign. This "education" of the immune system helps treat the patient because pancreatic cancer cells already present in a treated patient are believed to show some of the same differences from normal tissue as the modified pancreatic cancer cells in the product. Due to these similarities, the immune system, once "educated" by the Algenpantucel-L immunotherapy, identifies the patient's cancer as foreign and attacks.

The chemotherapy combination to be used in this study has been shown to improve survival in advanced pancreatic cancer and is being combined with an experimental pancreatic cancer immunotherapy that stimulates the immune system to recognize and attack the cancer. One goal of this study is to determine whether chemotherapy and immunotherapies can work cooperatively to increase anti-tumor effects to levels beyond what would be seen with either treatment alone.

In this experimental study, all patients are given a strong combination of anti-tumor chemotherapies while some patients are also given injections of an immunotherapy drug consisting of two types of pancreatic cancer cells that we have modified to make them more easily recognized and attacked by the immune system. We propose to test this new treatment protocol in patients with locally advanced pancreatic cancer to demonstrate that treatment with the immunotherapy increases the time until the tumor progresses or increases overall survival when given in combination with the current standard of care therapy for this disease.

DETAILED DESCRIPTION:
This protocol attempts to treat pancreatic cancer therapy using a naturally occurring barrier to xenotransplantation in humans to increase the efficacy of immunizing patients against their pancreatic cancer. In this protocol, the transfer of the murine α(1,3) galactosyltransferase [α(1,3)GT] gene to immunotherapy component cells results in the cell surface expression of α(1,3)galactosyl-epitopes (αgal) epitopes on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response. This response occurs when organs are transplanted from lower animal donor species into primates and results in rapid destruction of transplanted tissue and an augmented response against transplant antigens, including antigens not related to the αgal epitopes. Human hosts have pre-existing anti-α-gal antibodies that are thought to result from chronic immunological stimulation due to exposure to α-gal epitopes that are naturally expressed on normal gut flora and these antibodies may comprise up to 1% of serum immunoglobulin G (IgG). Opsonization and lysis of the immunotherapy component cells mediated by this antibody is believed to increase the efficiency of antigen processing by targeting vaccine components to antigen presenting cells via the Fcγ receptor.

ELIGIBILITY:
Inclusion Criteria:

* A histological diagnosis of adenocarcinoma of the pancreas confirmed by pathology.
* Patients must have borderline resectable or locally advanced unresectable pancreatic cancer with no metastatic spread as determined by a baseline diagnostic CT scan with intravenous contrast (or MRI). CT should be performed according to a defined pancreas protocol such as triphasic cross-sectional imaging with thin slices. Optimal multi-phase technique including a non-contrast phase plus arterial, pancreatic parenchymal and portal venous phase of contrast enhancement with thin cuts (3mm) throughout the abdomen is preferred. Studies must be evaluated by a radiologist and/or surgeon and deemed borderline resectable or locally advanced unresectable as defined per the NCCN Practice Guidelines in Oncology V2.2012, as:
* Borderline resectable- Tumors considered borderline resectable are defined as follows:

  1. No distant metastases
  2. Venous involvement of the SMV/portal vein demonstrating tumor abutment with impingement and narrowing of the lumen, encasement of the SMV/portal vein but without encasement of the nearby arteries, or short-segment venous occlusion resulting from either tumor thrombus or encasement but with suitable vessel proximal and distal to the area of vessel involvement, allowing for safe resection and reconstruction
  3. Gastroduodenal artery encasement up to the hepatic artery with either short segment encasement or direct abutment of the hepatic artery without extension to the celiac axis.
  4. Tumor abutment of the SMA not to exceed greater than 180 degrees of the circumference of the vessel wall.
* Tumors considered to be unresectable due to local advancement include an absence of distant metastases as well as:

  1. Head: Greater than 180 degrees SMA encasement or any celiac abutment or unreconstructible SMV/portal occlusion or aortic invasion or encasement.
  2. Body: Greater than 180 degrees SMA or celiac encasement or unreconstructible SMV/portal occlusion or aortic invasion.
  3. Tail: SMA or celiac encasement greater than 180 degrees.
  4. Nodal status: Involvement of lymph nodes beyond the field of resection should be considered unresectable due to distant spread and therefore not eligible for this protocol.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Serum albumin ≥ 2.0 gm/dL.
* Expected survival ≥ 6 months.
* Adequate organ function including:

  1. Marrow: WBC ≥3000/mm^3 and platelets ≥100,000/mm^3.
  2. Hepatic: serum total bilirubin ≤ 1.5 mg/dL, ALT (SGPT) and AST (SGOT) ≤3 x upper limit of normal (ULN) at time of enrollment. If a patient has elevated liver function tests at the time of initial presentation or develops them during work-up and they are the result of a mechanical obstruction of biliary drainage by tumor compression or invasion, a biliary drain may be placed as described in NCCN Practice Guidelines in Oncology V2.2012. If drainage allows for the liver function tests to come within inclusion criteria, the patient may be enrolled.
  3. Renal: serum creatinine (sCr) ≤2.0 x ULN, or creatinine clearance (Ccr) ≥30 mL/min.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* All subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental product, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active metastases.
* Other malignancy within five years, unless the probability of recurrence of the prior malignancy is <5% as determined by the Principal Investigator based on available information. Patient's curatively treated for squamous and basal cell carcinoma of the skin or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant.
* Current, active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking chronic systemic corticosteroid therapy for any reason are not eligible. Subjects may receive steroids as prophylactic anti-emetics per the FOLFIRINOX or gemcitabine/nab-paclitaxel regimen. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require chronic systemic corticosteroids after beginning treatment, will be removed from study.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias within the last six months.
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., active liver cirrhosis) or a serious illness in medical opinion of the clinical investigator.
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* A known history of allergy or hypersensitivity to any of the study drugs or any of their excipients.
* Pregnant or nursing women due to the unknown effects of immunization on the developing fetus or newborn infant. (For patients with child bearing potential, a βHCG must be completed within 14 days of first treatment).
* Known HIV positive.
* Prior treatment with chemotherapy or radiation for pancreatic cancer or prior treatment with radiation for other diagnoses to expected pancreatic cancer treatment fields.
* Current grade II or higher peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07-29 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 13.5 months (assuming enrollment period of 1-2 years)
  The primary objective of this study is to assess overall survival (OS) in pancreatic cancer patients with borderline resectable or locally advanced unresectable pancreatic cancer who will receive a regimen of FOLFIRINOX or gemcitabine/nab-paclitaxel with or without algenpantucel-L Immunotherapy.

SECONDARY OUTCOMES:
Progression Free Survival | 13.5 months (assuming enrollment period of 1-2 years)
  A secondary objective of this study is to assess progression free survival after treatment with a regimen of FOLFIRINOX or gemcitabine/nab-paclitaxel with or without algenpantucel-L immunotherapy in subjects who have borderline resectable or locally advanced pancreatic cancer.
Frequency and grade of adverse events of FOLFIRINOX or gemcitabine/nab-paclitaxel in combination with algenpantucel-L Immunotherapy versus FOLFIRINOX or gemcitabine/nab-paclitaxel alone | 13.5 months (assuming enrollment period of 1-2 years)
  A secondary objective of this study is to assess the safety (frequency and grade of adverse events) of administration of algenpantucel-L Immunotherapy given in combination with a standard of care regimen of chemotherapy (FOLFIRINOX or gemcitabine/nab-paclitaxel, to be referred to as standard of care, or SOC).
Immune Response | 13.5 months (assuming enrollment period of 1-2 years)
  A secondary objective of this study is to assess the immunologic responses of subjects with pancreatic cancer undergoing antitumor immunization with algenpantucel-L Immunotherapy as measured by correlative laboratory studies.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Institute for Medical Research, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Stamford Hospital, Stamford, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - USF Tampa General, Tampa, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville, Louisville, Kentucky
  - Beaumont CCOP, Royal Oak, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Renown Regional Medical Center, Reno, Nevada
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington - Seattle Cancer Center Alliance, Seattle, Washington
  - Vince Lombardi Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Hewitt DB, Nissen N, Hatoum H, Musher B, Seng J, Coveler AL, Al-Rajabi R, Yeo CJ, Leiby B, Banks J, Balducci L, Vaccaro G, LoConte N, George TJ, Brenner W, Elquza E, Vahanian N, Rossi G, Kennedy E, Link C, Lavu H. A Phase 3 Randomized Clinical Trial of Chemotherapy With or Without Algenpantucel-L (HyperAcute-Pancreas) Immunotherapy in Subjects With Borderline Resectable or Locally Advanced Unresectable Pancreatic Cancer. Ann Surg. 2022 Jan 1;275(1):45-53. doi: 10.1097/SLA.0000000000004669. PMID 33630475